CLINICAL TRIAL: NCT07223619
Title: PILOT Study: Treatment of Borderline Personality Disorder by Targeting Ventrolateral Prefrontal-amygdala Circuit With Network-based Neuronavigated Transcranial Magnetic Stimulation
Brief Title: PILOT Phase: BPD Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-1207
Record Dates: First submitted 2025-10-27; First posted 2025-11-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder
Keywords: BPD; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stimulation to Ventrolateral Prefrontal Cortex (Experimental): Each subjects will receive Transcranial Magnetic Stimulation or TMS to 3 different brain regions in 3 separate study visits spaced by at least 4 days (order randomized and counterbalanced amongst subjects).
  1. Right Ventrolateral Prefrontal Cortex or VLPFC
  2. Left VLPFC
  3. Bilateral: left and right VLPFC within 1 session
  The experimenters will utilize the MagVenture MagPro X100 stimulator equipped with the Cool B70 coil stimulate The TMS protocol includes 1800 pulses of excitatory intermittent theta burst stimulation (iTBS) at 120% MT intensity. This protocol will take less than 9 minutes (for each target).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain to improve symptoms of depression. Using pulsed magnetic fields, transcranial magnetic stimulation therapy stimulates the part of the brain thought to be involved with mood regulation. These magnetic fields do not directly affect the whole brain; they only reach about 2-3 centimeters into the brain directly beneath the treatment coil.As these magnetic fields move into the brain, they produce very small electrical currents. These electrical currents activate cells within the brain, causing them to rewire, a process called neuroplasticity.

SUMMARY:
This pilot study aims to identify the area of the brain best suited for the treatment of Borderline Personality disorder (BPD). The study investigators will test whether repetitiveTranscranial Magnetic Stimulation (rTMS), a gentle non-invasive brain stimulation method, can improve regulation of emotions and impulsivity in individuals with BPD.

This study will enroll up to 20 participants. Participant will be consented for the study remotely via a secure internet platform called Zoom. Participants will undergo 1 Magnetic Resonance Imaging or MRI scan and up to 3 brain stimulation of transcranial magnetic stimulation or TMS sessions, and cognitive behavioral testing on a computer.

Participants will complete 4 in-person visits over the course of up to 3 weeks.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a serious neuropsychiatric illness with a prevalence of 1-5% in the general population. Two core symptoms of BPD are emotional dysregulation and increased impulsivity. These dysfunctions are associated with depression, anxiety, and impulsive acts, particularly acts of self-harm that may include suicide. Current treatment options for BPD include specialized psychotherapies and pharmacotherapy, which are of limited beneﬁt for many patients. There is an urgent need for development of novel and more eﬀective treatments.

BPD may arise from dysfunction of brain circuits involved in emotional regulation. A circuit-based treatment such as repetitive Transcranial Magnetic Stimulation (rTMS) holds promise for treatment of BPD. Several recent studies examined rTMS treatment in BPD and found it was well tolerated with encouraging signs of clinical eﬃcacy. Advances in aﬀective neuroscience, combined with progress in brain imaging and neuromodulation technology, make it possible to develop new circuit-based approaches to rTMS that could enhance eﬃcacy for treatment for BPD. Evidence from task- based neuroimaging in BPD showed hyperactivity in the amygdala (a brain structure implicated in the generation of negative emotions) along with diminished top-down prefrontal-amygdala circuit control. These ﬁndings suggest that neuroimaging-guided rTMS stimulation of this circuit could enhance emotional regulation and behavioral control in patients with BPD and have greater therapeutic beneﬁt.

This project aims to explore a novel circuit-based rTMS treatment protocol for BPD. 20 subjects with BPD will be recruited and undergo resting-state functional Magnetic Resonance Imaging (fMRI) to identify regions in the right and left ventrolateral prefrontal cortex (VLPFC) having strongest connectivity with the right and left amygdala. These will be used as individualized targets for neuronavigated excitatory intermittent theta burst (iTBS) rTMS of right, left, and bilateral VLPFC. Change in measures of impulse control and emotion regulation will be examined pre-post single rTMS sessions to determine which stimulation target(s) show the greatest VLPFC-amygdala circuit engagement.

The study investigators will examine the eﬀects of right-sided, left-sided, and bilateral VLPFC stimulation in 20 subjects to determine which target(s) show the greatest signal of engagement of the VLPFC-amygdala network.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-65
* DSM-5 Diagnosis of Borderline Personality Disorder (BPD) based upon a psychiatric evaluation and ZAN-BPD scale
* Fluent English speaker
* Ability to give informed consent

Exclusion Criteria:

* Medical conditions that prevent TMS or MRI to be performed safely upon evaluation by the study psychiatrist
* Active alcohol or drug abuse of such severity that it would pose a risk for TMS administration (i.e., unstable motor thresholds or increased risk for seizure)
* Active suicidal plan
* Current diagnosis of Psychotic or Bipolar disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Delay Discounting Task (Odum, 2011) | Baseline, Visit 4 (up to 3 weeks)
  The Delay Discounting Task (DDT) is cognitive behavioral task performed to evaluate how individuals value rewards over time. It measures the tendency of individuals to prefer smaller, immediate rewards over larger, delayed ones. This behavior is known as delay discounting.
Cognitive Reappraisal of Social Exclusion Pain Task (Zhao et al., 2021) | Baseline, Visit 4 (up to 3 weeks)
  This task involves a comparison between a social exclusion group and a social inclusion group, and uses a pain-induction or pain-stimulus paradigm to measure the effects of social exclusion on individuals' perception and regulation of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Semel Institute/ UCLA TMS, Los Angeles, California, United States